CLINICAL TRIAL: NCT01251562
Title: A Phase 1 Dose Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of Sterile Compound c31510 for Injection Administered Intravenously to Subjects With Solid Tumors
Brief Title: Safety Study of Sterile Compound C31510 for Injection to Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BPGbio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTL0510
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2019-07

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Cohort 1 (Experimental): 5.62 mg/kg
  Sterile Compound C31510 for Injection
  Interventions: Drug: Sterile Compound C31510 for Injection
- Cohort 2 (Experimental): 11.25 mg/kg
  Sterile Compound C31510 for Injection
  Interventions: Drug: Sterile Compound C31510 for Injection
- Cohort 3 (Experimental): 22.5 mg/kg
  Sterile Compound C31510 for Injection
  Interventions: Drug: Sterile Compound C31510 for Injection
- Cohort 4 (Experimental): 33.0 mg/kg
  Interventions: Drug: Sterile Compound C31510 for Injection
- Cohort 5 (Experimental): 44.0 mg/kg
  Sterile Compound C31510 for Injection
  Interventions: Drug: Sterile Compound C31510 for Injection
- Cohort 6 (Experimental): 58.7 mg/kg
  Sterile Compound C31510 for Injection
  Interventions: Drug: Sterile Compound C31510 for Injection
- Cohort 7 (Experimental): 78.2 mg/kg
  Sterile Compound C31510 for Injection
  Interventions: Drug: Sterile Compound C31510 for Injection
- Cohort 8 (Experimental): 104.3 mg/kg
  Sterile Compound C31510 for Injection
  Interventions: Drug: Sterile Compound C31510 for Injection
- Cohort 9 (Experimental): 139.0 mg/kg
  Sterile Compound C31510 for Injection
  Interventions: Drug: Sterile Compound C31510 for Injection

INTERVENTIONS:
Drug: Sterile Compound C31510 for Injection — During the treatment period, subjects in each initial dose level cohort will have a single 4-hour IV infusion of C31510 at the assigned dose level of their particular cohort, three times per week for 26 days (on Day 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24 and 26) followed by a 28-day follow up period that will be counted from the first dose given on Day 1. In the absence of unacceptable toxicity or disease progression during the treatment period, those subjects may receive similar 28-day repeat treatment cycles of 3 times per week for up to 1 year, at the discretion of the investigator.

SUMMARY:
The primary objective of this clinical study is as follows:

• To determine the MTD and to assess the safety and tolerability of C31510 administered as a single 4-hour IV infusion (up to nine different dosages) in subjects with solid tumors

The secondary objective of this study is as follows:

• To evaluate plasma PK and estimate renal elimination of C31510 administered as a single 4-hour IV infusion (up to nine different dosages) in subjects with solid tumors

The exploratory objectives of this study are as follows:

* To evaluate the pharmacodynamic correlates of C31510 activity in plasma and peripheral blood cells
* To radiographically evaluate the effects of C31510 on tumors. In selected subjects, the effects on vascular permeability will be assessed by digital contrast enhanced (DCE)-magnetic resonance imaging (MRI)
* To evaluate tumor response (preliminary antitumor activity) after repeat administration of C31510
* Long-term safety and tolerability of C31510 after repeat administration

ELIGIBILITY:
Inclusion Criteria:

* The subject has a histologically confirmed solid tumor that is metastatic or unresectable for which standard curative measures do not exist or are no longer effective.
* The subject is at least 18 years old.
* The subject has an ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2.
* The subject has a life expectancy of greater than 3 months.
* The subject has organ and marrow function as follows: ANC>1500mm3, platelets>100,000 dl, hemoglobin >9 g/dL, bilirubin ≤ 1.5mg/dL, serum creatinine ≤1.5mg/dL or creatinine clearance >60 mL/min, and alanine aminotransferase (ALT), aspartate transaminase (AST) ≤2.5 times the upper limit of normal if no liver involvement or ≤5 times the upper limit of normal with liver involvement.
* The subject is capable of understanding and complying with the protocol and has signed the informed consent document.
* Sexually active subjects must use an accepted method of contraception during the course of the study.
* Female patients of childbearing potential must have a negative pregnancy test at enrollment.
* If a subject has received more than three prior regimens of cytotoxic chemotherapy, or more than two biological regimens, or more than 3000cGy to areas containing substantial marrow, the cohort review committee (CRC) must determine subject suitability prior to enrollment.

Exclusion Criteria:

* The subject has received chemotherapy or radiotherapy within 4 weeks or has received nitrosoureas or mitomycin C within 6 weeks prior to entering the study.
* The subject has received anti-angiogenesis drugs within 4 weeks prior to entering the study.
* The subject has received radiation to ≥25% of his or her bone marrow within 4 weeks of C31510IV treatment.
* The subject has received an investigational drug within 30 days of the first dose of study drug. 6 of 72
* The subject has not recovered to grade ≤1 from adverse events( AEs) due to investigational drugs or other medications, which were administered more than 4 weeks prior to study enrollment.
* The subject has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* The subject is pregnant or lactating.
* The subject is known to be positive for the human immunodeficiency virus (HIV)
* The subject has an inability or unwillingness to abide by the study protocol or cooperate fully with the investigator or designee.
* Must have not taken Vitamin D3 supplements in the last 30 days
* The subject is on HMG-CoA Reductase Inhibitors
* The subject is receiving digoxin, digitoxin, lanatoside C or any type of digitalis alkaloids
* The subject is receiving Colony Stimulating factors. The use of Colony Stimulating factors isf prohibited during the monitoring of DLT in this study.
* The subject is receiving Warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Tumor Assessment | at baseline and then once every two treatment cycles of 28 days (2 months) thereafter in the absence of clinical rapid progression of disease.
  Tumors will be assessed by standard methods ex. computerized tomography (CT), MRI etc; at baseline and then once every two treatment cycles of 28 days (2 months) thereafter in the absence of clinical rapid progression of disease.
  Assessment of tumor vascularity (using DCE-MRI) for at least 6 subjects who received C31510 at the MTD, will be done within 24 hours pre-dose and post-dose.

SECONDARY OUTCOMES:
blood samples taken for plasma pharmacokinetics (PK) evaluation | Blood samples collected at pre-dose, post-start of infusion at 0.5, 1, 2, 3.75 (15 min prior to end of infusion), 4.083 (5 min after the end of the infusion) 4.5, 6, 8, 10, and 24 hrs. after the start of the infusion
  samples are taken to evaluate plasma pharmacokinetics (PK) and estimate renal elimination of C31510 administered as a single IV infusion in subjects with solid tumors
  PK will be collected during Day 1 of the first month of each cohort at the following timepoints: pre-dose, post-start of infusion at 0.5, 1, 2, 3.75 (15 min prior to end of infusion), 4.083 (5 min after end of the infusion) 4.5, 6, 8, 10, and 24 hrs. after start of the infusion
  Additional PK will be done at pre-dose time and at 24 hours post the dose of Day 3, and on Day 28.
blood samples taken for plasma pharmacodynamics evaluation | Pharmacodynamic blood samples will be collected pre-dose and at 4 and 24 hours post dose after start of the infusion of Day 1 of each treatment cycle.
  blood samples are taken to evaluate the pharmacodynamic correlation of C31510 activity in plasma and peripheral blood cells

CONTACTS AND LOCATIONS:
Locations (1):
- Sarcoma Oncology Center, Santa Monica, California, United States